CLINICAL TRIAL: NCT04016350
Title: Impact of Moderate Intensity Exercise Training Combined With Inulin Propionate Ester Supplementation on Whole Body Resting Fat Oxidation and Body Weigh in Overweight Women
Brief Title: Impact of Exercise Combined With Inulin Propionate Ester on Fat Oxidation
Acronym: IPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UGlasgow IPE; BB/L004259/1 (Other Grant/Funding Number: BBSRC)
Record Dates: First submitted 2019-07-05; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Exercise; Inulin Propionate Ester
Keywords: Exercise,; Inulin Propionate Ester; Gut hormones; Body weigh; Fat oxidation; Overweight women
MeSH Terms: conditions — Motor Activity | interventions — Exercise; inulin-propionate ester

STUDY DESIGN:
Intervention Model Description: This is a randomised study with parallel design. Study participants underwent 4 week supervised moderate intensity exercise training combined either with IPE or cellulose as placebo supplementation at doses of 10g/day. Measurements were done before and after intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training with Inulin Propionate Ester (Experimental): Study participants underwent 4 week supervised moderate intensity exercise training combined with Inulin Propionate Ester supplementation at doses of 10g / day.
  Interventions: Behavioral: Exercise training with Inulin Propionate Ester
- Exercise Training with Placebo (Experimental): Study participants underwent 4 week supervised moderate intensity exercise training combined with cellulose as placebo at doses of 10g / day.
  Interventions: Behavioral: Exercise training with placebo

INTERVENTIONS:
Behavioral: Exercise training with Inulin Propionate Ester — Supervised moderate intensity exercise training combined with Inulin Propionate Ester supplementation conducted for 4 weeks.
  Arms: Exercise Training with Inulin Propionate Ester
Behavioral: Exercise training with placebo — Supervised moderate intensity exercise training combined with placebo conducted for 4 weeks
  Arms: Exercise Training with Placebo

SUMMARY:
There is evidence to suggest that responsiveness to exercise training programmes can be expected to be influenced by changes in resting fat oxidation, an important factor in the aetiology of obesity. Our previous work has shown that oral supplementation with inulin propionate ester (IPE) reduces intra-abdominal fat and prevents weight gain and that oral propionate intake enhances resting fat oxidation. The effects of IPE combined with exercise training on resting fat oxidation and body fatness are unknown. The aim of this study was to investigate the impact of 4-weeks IPE supplementation, in combination with a moderate intensity exercise training programme, on whole body fat oxidation and on plasma GLP-1 and PYY.

DETAILED DESCRIPTION:
Participants: Healthy overweight females with BMI >25 kg/m2 and 25-45 years of age were recruited through advertisements and word of mouth on the campus of the University of Glasgow or from other public places. Participants were required to be sedentary, non-smokers, with stable body weight for two months prior to the study enrollment, not pregnant, free of medication, nutritional supplementation or following any specific diet and with no antibiotic use for the past three months. Participants with chronic illness, eating disorders and history of gastrointestinal operations were excluded.

Study Design: This is a randomized study with a parallel design. Study participants underwent 4 week supervised moderate intensity exercise training combined either with IPE (EX/IPE) or cellulose as placebo (EX/Placebo) supplementation at doses of 10g / day. Supplements were provided as sachets containing white powder and participants were asked to consume one sachet per day with breakfast in a way convenient for each participant. Before the start of the study and at the end of the 4-week intervention, participants were asked to conduct a submaximal exercise test. Prior to the first and after the second submaximal exercise test, participants of both groups conducted a 7-hour experimental trial which involved collection of expired air and blood samples in fasted and postprandial states. Body weight and body composition were measured in the fasted state. Prior to the first 7-hour experimental trial, participants were asked to record their diet for 3 days and replicate this intake prior to the second 7-hour experimental trial.

ELIGIBILITY:
Inclusion Criteria:

Healthy, sedentary and overweight females with BMI >25 kg/m2 and stable body weight for two months prior to the study.

Exclusion Criteria:

Acute or chronic illness, eating disorders, history of gastrointestinal operations, smoking, pregnancy, taking supplements, and being on specific diet for the past three months.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-06-11 (Actual)

PRIMARY OUTCOMES:
Resting fat oxidation | 4 weeks
  Changes in resting fat oxidation measured in the fasted and postprandial states by means of indirect calorimetry (Oxycon Pro, Germany).
Resting carbohydrate oxidation | 4 weeks
  Changes in resting fat oxidation measured in the fasted and postprandial states by means of indirect calorimetry (Oxycon Pro, Germany).
Metabolic rate | 4 weeks
  Changes in resting energy expenditure measured in the fasted and postprandial states by means of indirect calorimetry (Oxycon Pro, Germany).

SECONDARY OUTCOMES:
Body weight | 4 weeks
  Changes in body weight measured by TANITA scales (TBF-300).
Body fat (%) | 4 weeks
  Changes in body fat expressed as percentage (proportion of fat to the total body weight) measured by TANITA scales (TBF-300).
Maximal oxygen consumption [Time Frame: 4 weeks] | 4 weeks
  Changes in maximal oxygen consumption (ml/kg/min) measured by Servomex Gas Analyser.
Peptide YY (PYY) | 4 weeks
  Changes in plasma concentration of fasting and postprandial PYY measured using ELISA (Merc Millipore) kit.
Glucagon-like peptide-1 (GLP-1) | 4 weeks
  Changes in plasma concentration of fasting and postprandial GLP-1 measured using ELISA (Merc Millipore) kit.
Height | 4 weeks
  Height (meters)measured by stadiometer, a vertical ruler with a sliding horizontal paddle which is adjusted to rest on the top of the head.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Morrison, PhD, Principal Investigator — University of Glasgow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malkova D, Polyviou T, Rizou E, Gerasimidis K, Chambers ES, Preston T, Tedford MC, Frost G, Morrison DJ. Moderate intensity exercise training combined with inulin-propionate ester supplementation increases whole body resting fat oxidation in overweight women. Metabolism. 2020 Mar;104:154043. doi: 10.1016/j.metabol.2019.154043. Epub 2019 Nov 29. PMID 31790692